CLINICAL TRIAL: NCT04952753
Title: An Open-label, Multi-center, ph II Platform Study Evaluating the Efficacy and Safety of NIS793 and Other New Investigational Drug Combinations With SOC Anti-cancer Therapy for the 2L Treatment of Metastatic Colorectal Cancer (mCRC)
Brief Title: Study of NIS793 and Other Novel Investigational Combinations With SOC Anti-cancer Therapy for the 2L Treatment of mCRC
Acronym: daNIS-3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to the halt of NIS793 treatment and urgent safety measures issued in July and August 2023, respectively, as continued evaluation of Standard of Care alone will not support the trial's purpose.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIS793E12201; 2021-000553-40 (EudraCT Number)
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: NIS793; metastatic colorectal cancer; colorectal cancer; transforming growth factor βeta (TGF-β); anti PD-1 monoclonal antibody
MeSH Terms: conditions — Colorectal Neoplasms | interventions — NIS-793; Bevacizumab; IFL protocol; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety run-in: NIS793+SOC (Investigational arm 1) (Experimental): In the safety run-in part for investigational arm 1, participants will be treated with a combination of SOC anti-cancer therapy (bevacizumab with either modified FOLFOX6 or FOLFIRI) and NIS793 to confirm the RP2D of the NIS793
  Interventions: Drug: NIS793; Drug: Bevacizumab; Drug: Modified FOLFOX6; Drug: FOLFIRI
- Expansion: NIS793+SOC (Investigational arm 1) (Experimental): In the expansion part, participants in the investigational arm 1 will be treated with a combination of SOC anti-cancer therapy (bevacizumab with either modified FOLFOX6 or FOLFIRI) and NIS793 at the RP2D defined in the safety run-in
  Interventions: Drug: NIS793; Drug: Bevacizumab; Drug: Modified FOLFOX6; Drug: FOLFIRI
- Expansion: SOC (control arm) (Active Comparator): In the expansion part, participants in the control arm will be treated with a combination of SOC anti-cancer therapy (bevacizumab with either modified FOLFOX6 or FOLFIRI)
  Interventions: Drug: Bevacizumab; Drug: Modified FOLFOX6; Drug: FOLFIRI
- Safety run-in: NIS793+Tislelizumab+SOC (Investigational arm 2) (Experimental): In the safety run-in part for investigational arm 2, participants will be treated with a combination of SOC anti-cancer therapy (bevacizumab with either modified FOLFOX6 or FOLFIRI), NIS793 and tislelizumab to confirm the RP2D of NIS793.
  Interventions: Drug: NIS793; Drug: Bevacizumab; Drug: Modified FOLFOX6; Drug: FOLFIRI; Drug: Tislelizumab
- Expansion: NIS793+Tislelizumab+SOC (Investigational arm 2) (Experimental): In the expansion part, participants in the investigational arm 2 will be treated with a combination of SOC anti-cancer therapy (bevacizumab with either modified FLOFOX6 or FOLFIRI) with NIS793 and tislelizumab at the RP2D for NIS793 defined in the safety run-in
  Interventions: Drug: NIS793; Drug: Bevacizumab; Drug: Modified FOLFOX6; Drug: FOLFIRI; Drug: Tislelizumab

INTERVENTIONS:
Drug: NIS793 — Investigational drug NIS793 will be administered intravenously (IV) at the dose and schedule determined in the safety run-in part.
  Arms: Expansion: NIS793+SOC (Investigational arm 1); Expansion: NIS793+Tislelizumab+SOC (Investigational arm 2); Safety run-in: NIS793+SOC (Investigational arm 1); Safety run-in: NIS793+Tislelizumab+SOC (Investigational arm 2)
Drug: Bevacizumab — Bevacizumab will be administered IV
Drug: Modified FOLFOX6 — 5-fluorouracil [continuous infusion], leucovorin [administered IV] (or levoleucovorin [administered IV]), and oxaliplatin [administered IV]
  Other Names: 5FU+Leucovorin+Oxaliplatin
Drug: FOLFIRI — 5-fluorouracil [continuous infusion], leucovorin [administered IV] (or levoleucovorin [administered IV]), and irinotecan [administered IV]
  Other Names: 5FU+Leucovorin+Irinotecan
Drug: Tislelizumab — Investigational drug tislelizumab will be administered intravenously (IV).
  Other Names: VDT482
  Arms: Expansion: NIS793+Tislelizumab+SOC (Investigational arm 2); Safety run-in: NIS793+Tislelizumab+SOC (Investigational arm 2)

SUMMARY:
The purpose of this study is to evaluate the preliminary efficacy and safety of NIS793 and other novel investigational combinations with standard of care (SOC) anti-cancer therapy vs SOC anti-cancer therapy for the second line treatment of mCRC.

This study aims to explore whether different mechanisms of action may reverse resistance and improve responsiveness to the currently considered SOC anti-cancer therapy in the second line metastatic colorectal cancer (mCRC) setting.

DETAILED DESCRIPTION:
This is an open-label, multi-center, phase II, 2-part platform study with Safety run-in and Expansion parts.

The platform design of this study is adaptive to allow flexibility in the introduction of additional treatment arms with new investigational drugs in combination with SOC anti-cancer therapy for the second line treatment of mCRC.

The study will include a control arm that will enroll participants treated with SOC anti-cancer therapy (bevacizumab with mFOLFOX6 or FOLFIRI) for the second line treatment of mCRC. The choice of the chemotherapy medications (mFOLFOX6 or FOLFIRI) will be determined by the Investigator based on prior exposure to oxaliplatin or irinotecan.

Each investigational arm will include a combination of an investigational drug and the SOC anti-cancer therapy. The first investigational arm of the study will explore the combination of anti-transforming growth factor β (TGF-β) monoclonal antibody, NIS793 with SOC anti-cancer therapy. The second investigational arm of the study will explore the combination of anti-transforming growth factor β (TGF-β) monoclonal antibody, NIS793 with Tislelizumab, which is an anti-PD1 monoclonal antibody, and SOC anti-cancer therapy. Combination of other investigational drugs with SOC anti-cancer therapy may be added by protocol amendments an additional investigational arms.

In each investigational arm, a Safety run-in part will be conducted before opening the expansion part to confirm the recommended phase 2 dose (RP2D) for a combination of any investigational drug with SOC anti-cancer therapy unless the dose has been confirmed externally to this trial.

The decision to open the Expansion part of the study will be based on dose confirmation of investigational drug with available safety, relevant PK and other relevant data from Safety run-in part. Participants in the expansion part will be randomized in 1:2 ratio to the control arm or investigational arm.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants age 18 or older with histologically or cytologically confirmed (by local laboratory and local clinical guidelines) metastatic colorectal adenocarcinoma that is not amenable to potentially curative surgery in the opinion of the investigator and progressed on or within 6 months after the last dose of one prior line of systemic anti-cancer therapy administered for metastatic disease.
* Presence of at least one measurable lesion assessed by CT and/or MRI according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Adequate organ function (assessed by central laboratory for eligibility).

Key Exclusion Criteria:

* Previously administered TGF-β targeted therapies or anti-cancer immunotherapy.
* Microsatellite instability-high (MSI-H)/mismatch repair-deficient (dMMR) and/or BRAFV600 mutation positive colorectal cancer.
* Known complete or partial dipyrimidine dehydrogenase (DPD) enzyme deficiency (testing for DPD enzyme deficiency is not mandatory unless required by local regulations and can be conducted at a local laboratory).
* For participants treated with irinotecan: Known history or clinical evidence of reduced UGT1A1 activity (testing for UGT1A1 status is not mandatory unless required by local regulations and can be conducted at a local laboratory).
* Participants who have not recovered from a major surgery performed prior to start of study treatment or have had a major surgery within 4 weeks prior to start of study treatment.
* Impaired cardiac function or clinically significant cardio-vascular disease.
* Participants with conditions that are considered to have a high risk of clinically significant gastrointestinal tract bleeding or any other condition associated with or history of significant bleeding.
* Stroke or transient ischemic attack, or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 3 months before start of study treatment.
* Pregnant or breast-feeding women.
* Women of childbearing potential, unless willing to use highly effective contraception methods during treatment and after stopping study treatments as required.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Safety run-in: Percentage of participants with dose limiting toxicities (DLTs) during the first cycle (4 weeks) of treatment. | Up to 4 weeks
  Percentage of participants with DLTs during the first cycle of treatment. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness or concomitant medication that occurs within the first cycle of treatment with NIS793 with or without tislelizumab in combination with Bevacizumab and modified FOLFOX6/ FOLFIRI and meets protocol defined DLT criteria.
Expansion: Progression-free survival (PFS) by investigator assessment per RECIST 1.1 | From randomization up to disease progression or death, assessed up to approximately 12 months
  PFS defined as the time from the date of enrollment (run-in part) or randomization (randomized part) to the date of the first documented progression based on investigator assessment and according to RECIST 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Safety run-in: Percentage of participants with Adverse Events (AEs) | Up to approximately 12 months
  Percentage of participants with AEs and SAEs including changes in laboratory parameters, vital signs, body weight and cardiac assessments
Safety run-in: Percentage of participants with dose interruptions and dose reductions of investigational drug | Upto approximately 12 months
  Tolerability measured by the percentage of subjects who have dose adjustments (interruptions or reductions) of investigational drug (e.g. NIS793, NIS793+tislelizumab)
Safety run-in: Dose intensity of investigational drug | Up to approximately 12 months
  Tolerability measured by the dose intensity of investigational drug (e.g. NIS793, NIS793+tislelizumab). Dose intensity will be computed as the ratio of actual cumulative dose received and actual duration of exposure
Safety run-in: PFS by investigator assessment per RECIST 1.1 | From enrollment up to disease progression or death, assessed up to approximately 12 months
  PFS defined as the time from the date of enrollment to the date of the first documented progression based on investigator assessment and according to RECIST 1.1 or death due to any cause.
Safety run-in: Overall response rate (ORR) by investigator assessment per RECIST 1.1 | Up to approximately 12 months
  ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per investigator assessment and according to RECIST 1.1
Safety run-in: Disease control rate (DCR) by investigator assessment per RECIST 1.1 | Up to approximately 12 months
  DCR is the proportion of participants with BOR of CR or PR or stable disease (SD) as per investigator assessment and according to RECIST 1.1
Safety run-in: Duration of response (DOR) by investigator assessment per RECIST 1.1 | From first documented response up to disease progression or death, assessed up to approximately 12 months
  DOR is defined as the duration of time between the date of the first documented response (CR or PR) and the date of first documented progression or death due to any cause
Safety run-in part: Overall Survival (OS) | From enrollment up to death, assessed up to approximately 12 months
  OS is defined as the time from the date of enrollment to date of death due to any cause.
Safety run-in: Time to response (TTR) by investigator assessment per RECIST 1.1 | From enrollment up to first documented response, assessed up to approximately 12 months
  TTR is defined as the duration of time between the date of enrollment and the date of first documented response of either CR or PR.
Expansion: Percentage of participants with Adverse Events (AEs) | Up to approximately 12 months
  Percentage of participants with AEs and SAEs including changes in laboratory parameters, vital signs, body weight and cardiac assessments
Expansion part: Percentage of participants with dose interruptions and dose reductions of investigational drug | Up to approximately 12 months
  Tolerability measured by the percentage of subjects who have dose adjustments (interruptions) of investigational drug (e.g. NIS793, NIS793+tislelizumab)
Expansion: Dose intensity of investigational drug | Up to approximately 12 months
  Tolerability measured by the dose intensity of investigational drug (e.g. NIS793, NIS793+Tislelizumab). Dose intensity will be computed as the ratio of actual cumulative dose received and actual duration of exposure
Expansion: Overall response rate (ORR) by investigator assessment per RECIST 1.1 | Up to approximately 12 months
  ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per investigator assessment and according to RECIST 1.1
Expansion: Disease control rate (DCR) by investigator assessment per RECIST 1.1 | Up to approximately 12 months
  DCR is the proportion of participants with BOR of CR or PR or stable disease (SD) as per investigator assessment and according to RECIST 1.1
Expansion: Duration of response (DOR) by investigator assessment per RECIST 1.1 | From first documented response up to disease progression or death, assessed up to approximately 12 months
  DOR is defined as the duration of time between the date of the first documented response (CR or PR) and the date of first documented progression or death due to any cause
Expansion part: Overall Survival (OS) | From randomization up to death, assessed up to approximately 12 months
  OS is defined as the time from the date of enrollment to date of death due to any cause.
Expansion: Time to response (TTR) by investigator assessment per RECIST 1.1 | From enrollment up to first documented response, assessed up to approximately 12 months
  TTR is defined as the duration of time between the date of enrollment and the date of first documented response of either CR or PR.
Maximum concentration (Cmax) of NIS793 | From the date of first study drug intake up to approximately 12 months
  Blood samples will be collected at indicated time-points for analysis of Cmax of NIS793
Maximum concentration (Cmax) of tislelizumab | From the date of first study drug intake up to approximately 12 months
  Blood samples will be collected at indicated time-points for analysis of Cmax of tislelizumab
Trough Concentration (Ctrough) of NIS793 | From the date of first study drug intake up to approximately 12 months
  Blood samples will be collected at indicated time-points for analysis of Ctrough of NIS793
Trough Concentration (Ctrough) tislelizumab | From the date of first study drug intake up to approximately 12 months
  Blood samples will be collected at indicated time-points for analysis of Ctrough of tislelizumab
Antidrug antibodies (ADA) at baseline | Baseline
  Prevalence of ADA (anti-NIS793, anti-tislelizumab) at baseline is defined as the proportion of participants who have an ADA positive result at baseline
ADA incidence on treatment | From the date of first study drug intake up to approximately 12 months
  Incidence of ADA (anti-NIS793, anti-tislelizumab) on treatment is defined as the proportion of participants who are treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (51):
- United States (7):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Michigan Medical, Ann Arbor, Michigan
  - WA Uni School Of Med, St Louis, Missouri
  - Astera Cancer Center, East Brunswick, New Jersey
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
- Australia (3):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Bendigo, Victoria
  - Novartis Investigative Site, Perth, Western Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (3):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- France (3):
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Nantes
- Germany (7):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ulm
- Hong Kong (2):
  - Novartis Investigative Site, Pokfulam
  - Novartis Investigative Site, Shatin
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Toyama
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- United Kingdom (3):
  - Novartis Investigative Site, Aberdeen, Grampian Region
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com